CLINICAL TRIAL: NCT03198065
Title: The Application of Minimally Invasive Single-incision Laparoscopic Surgery in Acute Abdomen
Brief Title: Single-incision Laparoscopic Surgery in Acute Abdomen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201702076RIND
Record Dates: First submitted 2017-06-18; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Acute Appendicitis
Keywords: Laparoscopic appendectomy; Single-incision laparoscopic appendectomy; Single-incision laparoscopic surgery setting; Simple appendicitis; Complicated appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-made glove setting (Experimental): The patients receive Hand-made glove setting
  Interventions: Procedure: Hand-made glove setting
- commercialized multiport setting (Experimental): The patients receive commercialized single-incision multiport setting
  Interventions: Procedure: Commercialized single-incision multiport setting

INTERVENTIONS:
Procedure: Hand-made glove setting — The patients receive Hand-made glove setting for single-incision laparoscopic appendectomy
  Arms: Hand-made glove setting
Procedure: Commercialized single-incision multiport setting — The patients receive commercialized single-incision multiport setting for single-incision laparoscopic appendectomy
  Arms: commercialized multiport setting

SUMMARY:
Since Semm et.al. reported the first case of laparoscopic appendectomy in 1983, minimally invasive surgery has become the main stay for treating of many surgical diseases. After the booming in the advancement of surgical instrument and breakthrough in surgical skills, the minimally invasive surgery has been widely applied to neurosurgery, spinal surgery, breast, thyroid, hernia surgery, etc. It has been proved that minimally invasive surgery is safe and effective, and further it achieves compatible results and outcomes in oncology and functional diseases. Minimally invasive surgery in alimentary tract, known as laparoscopic surgery, has been performed in gastric surgery (e.g. gastric cancer, tumor, functional disorders and bariatric surgery), hepatobiliary and pancreatic surgery (e.g. hepatectomy, cholecystectomy, and pancreatectomy), and colorectal surgery (e.g. colorectal cancer and functional bowel disease). Under a superior heritage of surgical skills from Taiwan university hospital, we introduced laparoscopic surgery in 1996 and currently, laparoscopic surgery becomes the mainstay of surgery in Yunlin branch. In 2015, there were 600 laparoscopic surgery in our hospital, while 150 colorectal laparoscopic surgery in the same year. In recent years, single-incisional laparoscopic surgery has emerged to become one of the focused topic in the world and seemly in our department. Through single-incision surgery, we attempted to minimize the incision wound to achieve better cosmesis and faster recovery. By the valuable clinical experiences gathering in our hospital (Yunlin branch) in recent 10 years, we contemplate two-step plans: first, by retrospective data collection, we can explain the clinical problems based on current statistical results. Second, based on prior (step 1) retrospective findings, a prospective study could be conducted for more evident results.

DETAILED DESCRIPTION:
The aim of this study is to compare two kinds of single-incision laparoscopic surgery setting including hand-made glove setting and commercialized single-incision multiport setting. The preoperative, intraoperative and postoperative data will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The patients admitted to the NTUH Yunlin branch diagnosed clinically as acute appendicitis
2. The patients with clinically suspected right lower quadrant pain and acute appendicitis could not be excluded

Exclusion Criteria:

1. Not eligible to underwent laparoscopic surgery because of compromised cardiopulmonary function or major laparotomy surgery
2. Decide to receive non-surgical treatment of the acute appendicitis
3. Age<20, or could not exercise the right of autonomy or unwilling to participate the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-17 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | around 2 years
  Postoperative pain is measured by visual pain scale
wound cosmesis | around 2 years
  The cosmesis is measure by the length of the incision

SECONDARY OUTCOMES:
Operative time | around 2 years
  By chart review
Visceral/vascular injuries | around 2 years
  Recorded on the operative note
Conversion | around 2 years
  Recorded on the operative note
Wound infection/surgical site infection | around 2 years
  By chart review
Intra-abdominal collection | around 2 years
  Defined by evidence on any image modalities
Postoperative ileus | around 2 years
  Defined by ileus physically or by image
Length of hospitalization | around 2 years
  By chart review
Time to return work | around 2 years
  By chart review

CONTACTS AND LOCATIONS:
Overall Officials: Peng-shen Lai, M.D., Study Director — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No